CLINICAL TRIAL: NCT01652651
Title: The Contribution of Risk and Resilience Factors in Learning Disabilities Population to Academic and Emotional Development
Brief Title: Risk and Resilience Factors in Learning Disabilities Population
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 5383
Record Dates: First submitted 2012-06-17; First posted 2012-07-30 (Estimated); Last update posted 2012-07-30 (Estimated); Status verified 2012-06

CONDITIONS: Learning Disorders
Keywords: Learning Disorders
MeSH Terms: conditions — Learning Disabilities

ARMS (1):
- Psychological Intervention (Experimental)
  Interventions: Behavioral: I Can Succeed ICS

INTERVENTIONS:
Behavioral: I Can Succeed ICS — ICS is a manual-based psychological intervention aimed to address both emotional and academic-executive functions aspects of LD.It consists of acute phase (13 once a week sessions) and follow-up phase (6 sessions over 18 months). ICS focuses on developing intrapersonal skills (e.g. self awareness, goal setting, organizational skills), interpersonal skills (e.g. communication, problem solving)and school/community skills (i.e. strengthening the family-school relationship) (Kopelman-Rubin et al., 2011).

SUMMARY:
The purpose of this study is to report preliminary outcomes of executive function and psychopathology symptoms of a manual-based psychological intervention for adolescents diagnosed with learning disorders- I can succeed (ICS).

ELIGIBILITY:
Inclusion Criteria:

* Learning Disorder diagnosis
* Normal range IQ
* Regular class attendance

Exclusion Criteria:

* Suicidal ideation and psychosis

Ages: 11 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2009-05; Primary Completion 2012-04 (Actual); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Change in Child Behavior Checklist (CBCL) (Achenbach, 1991). | base line (time 0) and end of treatment (3 month)
  The Child Behavior Checklist (CBCL) is a device by which parents and teachers rate a child's problem behaviors and competencies. It consists of 112 behavioral items (and 1 open-ended item) scored on a 3-step response scale from Not true (0) to Very true or Often true (2). Subscales include Aggressive Behavior, Anxious/Depressed, Attention Problems, Delinquent Rule-Breaking Behavior, Social Problems, Somatic Complaints, Thought Problems, Withdrawn, Externalizing, Internalizing, Total Problems, plus DSM-oriented scales.

SECONDARY OUTCOMES:
Change in The standardized Brain Resource cognition assessment, ''IntegNeuro,'' (Clark et al., 2006). | base line (time 0) and end of treatment (3 month)
  A computerized standardized assessment of Executive Functions and Continuous Performance Test

CONTACTS AND LOCATIONS:
Overall Officials: Daphne Kopelman-Rubin, Ph.D, Principal Investigator — Schneider's Children Medical Center of Israel
Locations (1):
- Schneider Children Medical Center of Israel, Petah Tikva, Israel